CLINICAL TRIAL: NCT03430167
Title: Supervised Physiotherapy Versus a Home Exercise Program After Reverse Total Shoulder Arthroplasty: a Randomized Clinical Trial
Brief Title: Reverse Shoulder Replacement: Formal vs. Home Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201703024
Record Dates: First submitted 2018-01-23; First posted 2018-02-12 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Arthropathy Associated With Other Conditions
Keywords: Reverse Total Shoulder Arthroplasty; post operative physical therapy
MeSH Terms: interventions — Home Infusion Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: post operative assessor obtaining range of motion and performing physical exam will be blinded to participant's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I - Formal Therapy (Other): Supervised physical therapy will be ordered 2 times/week initially for 6 weeks and then tailored to a minimum of 1 visit/week based upon the individual progress of each patient. Home exercises will be provided to the patient by the therapist to be performed daily. Supervised physical therapy will be discontinued once the patient demonstrates independence with the final phase of rehabilitation, which represents the graduated strengthening program.
  Interventions: Other: formal therapy
- Group II - Home Therapy (Other): In the study group all patients will be instructed in a standardized fashion regarding a home exercise program. This program will involve a standardized a set of five exercises. These exercises will be reviewed with patients in clinic in a standardized fashion and patients will be provided with an instructive hand-out.
  Interventions: Other: home therapy

INTERVENTIONS:
Other: home therapy — Patients will be given a set of instructions for completing home therapy for range of motion and strengthening
  Arms: Group II - Home Therapy
Other: formal therapy — Patients will be sent to physical therapist for formal treatment to regain range of motion and strengthening exercises
  Arms: Group I - Formal Therapy

SUMMARY:
The purpose of this study is to compare range of motion between a structured home exercise program to supervised physiotherapy post-operatively after Reverse Total Shoulder Replacement is performed for rotator cuff tear arthropathy/massive cuff tear through a single-center, assessor-blinded, randomized clinical trial.

DETAILED DESCRIPTION:
All patients who are evaluated by one of three Shoulder/Elbow Fellowship-trained surgeons at Washington University Department of Orthopedic Surgery and who meet the inclusion criteria will be offered enrollment in the study. Following consent the participant will be asked to undergo an exam of the shoulder and complete questionnaires related to shoulder pain and function.

Demographic information, health history related to the affected shoulder, and co-morbidity data will also be collected preoperatively.

Patients will be randomized to either a simple, standardized home exercise program or a supervised physiotherapy program administered by a physical therapist after undergoing a standardized operative protocol for reverse total shoulder arthroplasty.

Post-operative range of motion will be measured in a blinded fashion at 6 weeks, 3 months, 6 months, and 12 months. A blinded observer will simultaneously measure validated functional outcomes scores including the Western Ontario Osteoarthritis Score, American Shoulder and Elbow Surgeons Score and Visual Analogue Score for pain pre-operatively and at 6 weeks, 3 months, 6 months, and 12 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Primary RTSA for the diagnosis of rotator cuff tear arthropathy (RCTA) or irreparable rotator cuff tear.
2. A pre-operative plan for RTSA
3. Age >60

Exclusion Criteria:

1. Active infection
2. Incompetent deltoid muscle
3. Unwillingness or inability to participate in a home exercise program
4. Medically unfit for operative intervention
5. Revision RTSA
6. RTSA for glenohumeral osteoarthritis or proximal humerus fracture
7. Unwillingness to participate in the study
8. Inability to read or comprehend written instructions

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Range of Motion Outcomes | Baseline and at 6 weeks, 3 months, 12 months and 24 months post-operatively
  Compare change in shoulder range of motion after supervised physiotherapy versus a structured home exercise program after Reverse Total Shoulder Arthroplasty.

SECONDARY OUTCOMES:
Clinical Outcome Scores - Quality of Life | Baseline and at 6 weeks, 3 months, 12 months and 24 months post-operatively
  Compare change in The Western Ontario Osteoarthritis Score (WOOS) after supervised physiotherapy versus a structured home exercise program after Reverse Total Shoulder Arthroplasty.
  The WOOS includes 19 items (0-100 visual analog scale) which assess 1. pain and physical symptoms 2. sports, recreation, and work 3. lifestyle function, and 4. emotional function. A higher score represents a worse outcome.
Clinical Outcome Scores - Functional | Baseline and at 6 weeks, 3 months, 2 months and 24 months post-operatively
  Compare change in American Shoulder and Elbow Surgeons Score (ASES) after supervised physiotherapy versus a structured home exercise program after Reverse Total Shoulder Arthroplasty.
  The ASES includes 1 pain item (0-100 visual analog scale) and 10 items which assess functional status (0=Unable to do, 1=Very difficult to do, 2=Somewhat difficult, 3=Not difficult). A higher score represents a better outcome.
Clinical Outcome Scores - Pain | Baseline and at 6 weeks, 3 months, 12 months and 24 months post-operatively
  Compare change in Visual Analogue Pain Score (0-100) after supervised physiotherapy versus a structured home exercise program after Reverse Total Shoulder Arthroplasty.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Chamberlain, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- University of Utah - Orthopedics, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SH, Wise BL, Zhang Y, Szabo RM. Increasing incidence of shoulder arthroplasty in the United States. J Bone Joint Surg Am. 2011 Dec 21;93(24):2249-54. doi: 10.2106/JBJS.J.01994. PMID 22258770
- [Background] Schairer WW, Nwachukwu BU, Lyman S, Craig EV, Gulotta LV. National utilization of reverse total shoulder arthroplasty in the United States. J Shoulder Elbow Surg. 2015 Jan;24(1):91-7. doi: 10.1016/j.jse.2014.08.026. Epub 2014 Oct 29. PMID 25440519
- [Background] Lawrence TM, Ahmadi S, Sanchez-Sotelo J, Sperling JW, Cofield RH. Patient reported activities after reverse shoulder arthroplasty: part II. J Shoulder Elbow Surg. 2012 Nov;21(11):1464-9. doi: 10.1016/j.jse.2011.11.012. Epub 2012 Feb 22. PMID 22365817
- [Background] Young SW, Zhu M, Walker CG, Poon PC. Comparison of functional outcomes of reverse shoulder arthroplasty with those of hemiarthroplasty in the treatment of cuff-tear arthropathy: a matched-pair analysis. J Bone Joint Surg Am. 2013 May 15;95(10):910-5. doi: 10.2106/JBJS.L.00302. PMID 23677358
- [Background] Guery J, Favard L, Sirveaux F, Oudet D, Mole D, Walch G. Reverse total shoulder arthroplasty. Survivorship analysis of eighty replacements followed for five to ten years. J Bone Joint Surg Am. 2006 Aug;88(8):1742-7. doi: 10.2106/JBJS.E.00851. PMID 16882896
- [Background] Mulieri P, Dunning P, Klein S, Pupello D, Frankle M. Reverse shoulder arthroplasty for the treatment of irreparable rotator cuff tear without glenohumeral arthritis. J Bone Joint Surg Am. 2010 Nov 3;92(15):2544-56. doi: 10.2106/JBJS.I.00912. PMID 21048173
- [Background] Steen BM, Cabezas AF, Santoni BG, Hussey MM, Cusick MC, Kumar AG, Frankle MA. Outcome and value of reverse shoulder arthroplasty for treatment of glenohumeral osteoarthritis: a matched cohort. J Shoulder Elbow Surg. 2015 Sep;24(9):1433-41. doi: 10.1016/j.jse.2015.01.005. Epub 2015 Mar 11. PMID 25769903
- [Background] Wall B, Nove-Josserand L, O'Connor DP, Edwards TB, Walch G. Reverse total shoulder arthroplasty: a review of results according to etiology. J Bone Joint Surg Am. 2007 Jul;89(7):1476-85. doi: 10.2106/JBJS.F.00666. PMID 17606786
- [Background] Favard L, Levigne C, Nerot C, Gerber C, De Wilde L, Mole D. Reverse prostheses in arthropathies with cuff tear: are survivorship and function maintained over time? Clin Orthop Relat Res. 2011 Sep;469(9):2469-75. doi: 10.1007/s11999-011-1833-y. PMID 21384212
- [Background] Kiet TK, Feeley BT, Naimark M, Gajiu T, Hall SL, Chung TT, Ma CB. Outcomes after shoulder replacement: comparison between reverse and anatomic total shoulder arthroplasty. J Shoulder Elbow Surg. 2015 Feb;24(2):179-85. doi: 10.1016/j.jse.2014.06.039. Epub 2014 Sep 9. PMID 25213827
- [Background] Cazeneuve JF, Cristofari DJ. The reverse shoulder prosthesis in the treatment of fractures of the proximal humerus in the elderly. J Bone Joint Surg Br. 2010 Apr;92(4):535-9. doi: 10.1302/0301-620X.92B4.22450. PMID 20357330
- [Background] Levy JC, Badman B. Reverse shoulder prosthesis for acute four-part fracture: tuberosity fixation using a horseshoe graft. J Orthop Trauma. 2011 May;25(5):318-24. doi: 10.1097/BOT.0b013e3181f22088. PMID 21464740
- [Background] Frankle M, Siegal S, Pupello D, Saleem A, Mighell M, Vasey M. The Reverse Shoulder Prosthesis for glenohumeral arthritis associated with severe rotator cuff deficiency. A minimum two-year follow-up study of sixty patients. J Bone Joint Surg Am. 2005 Aug;87(8):1697-705. doi: 10.2106/JBJS.D.02813. PMID 16085607
- [Background] Chalmers PN, Slikker W 3rd, Mall NA, Gupta AK, Rahman Z, Enriquez D, Nicholson GP. Reverse total shoulder arthroplasty for acute proximal humeral fracture: comparison to open reduction-internal fixation and hemiarthroplasty. J Shoulder Elbow Surg. 2014 Feb;23(2):197-204. doi: 10.1016/j.jse.2013.07.044. Epub 2013 Sep 27. PMID 24076000
- [Background] Cvetanovich GL, Chalmers PN, Streit JJ, Romeo AA, Nicholson GP. Patients Undergoing Total Shoulder Arthroplasty on the Dominant Extremity Attain Greater Postoperative ROM. Clin Orthop Relat Res. 2015 Oct;473(10):3221-5. doi: 10.1007/s11999-015-4400-0. Epub 2015 Jun 12. PMID 26066068
- [Background] Levy JC, Everding NG, Gil CC Jr, Stephens S, Giveans MR. Speed of recovery after shoulder arthroplasty: a comparison of reverse and anatomic total shoulder arthroplasty. J Shoulder Elbow Surg. 2014 Dec;23(12):1872-1881. doi: 10.1016/j.jse.2014.04.014. Epub 2014 Jun 26. PMID 24981553
- [Background] Young AA, Smith MM, Bacle G, Moraga C, Walch G. Early results of reverse shoulder arthroplasty in patients with rheumatoid arthritis. J Bone Joint Surg Am. 2011 Oct 19;93(20):1915-23. doi: 10.2106/JBJS.J.00300. PMID 22012529
- [Background] Hattrup SJ, Sanchez-Sotelo J, Sperling JW, Cofield RH. Reverse shoulder replacement for patients with inflammatory arthritis. J Hand Surg Am. 2012 Sep;37(9):1888-94. doi: 10.1016/j.jhsa.2012.05.015. Epub 2012 Jun 30. PMID 22749484
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Charlson ME, Sax FL, MacKenzie CR, Braham RL, Fields SD, Douglas RG Jr. Morbidity during hospitalization: can we predict it? J Chronic Dis. 1987;40(7):705-12. doi: 10.1016/0021-9681(87)90107-x. PMID 3110198
- [Background] Walch G, Badet R, Boulahia A, Khoury A. Morphologic study of the glenoid in primary glenohumeral osteoarthritis. J Arthroplasty. 1999 Sep;14(6):756-60. doi: 10.1016/s0883-5403(99)90232-2. PMID 10512449
- [Background] Kappe T, Cakir B, Reichel H, Elsharkawi M. Reliability of radiologic classification for cuff tear arthropathy. J Shoulder Elbow Surg. 2011 Jun;20(4):543-7. doi: 10.1016/j.jse.2011.01.012. Epub 2011 Mar 30. PMID 21454101
- [Background] Sirveaux F, Favard L, Oudet D, Huquet D, Walch G, Mole D. Grammont inverted total shoulder arthroplasty in the treatment of glenohumeral osteoarthritis with massive rupture of the cuff. Results of a multicentre study of 80 shoulders. J Bone Joint Surg Br. 2004 Apr;86(3):388-95. doi: 10.1302/0301-620x.86b3.14024. PMID 15125127